CLINICAL TRIAL: NCT05183347
Title: Safety, Tolerability, and Pharmacokinetics of Single Rising Oral Doses and Multiple Oral Doses of BI 1291583 in Healthy Male Japanese Subjects (Double-blind, Randomised, Placebo-controlled, Parallel Group Design)
Brief Title: A Study in Healthy Japanese Men to Test How Well Different Doses of BI 1291583 Are Tolerated
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1397-0003
Record Dates: First submitted 2021-12-22; First posted 2022-01-10 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- SRD: Dose Group 1 (Experimental): SRD: single-rising dose
  Interventions: Drug: BI 1291583
- SRD: Dose Group 2 (Experimental): SRD: single-rising dose
  Interventions: Drug: BI 1291583
- SRD: Dose Group 3 (Experimental): SRD: single-rising dose
  Interventions: Drug: BI 1291583
- MD: Dose Group 4 (Experimental): MD: multiple doses
  Interventions: Drug: BI 1291583
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1291583 — BI 1291583
  Other Names: Verducatib
  Arms: MD: Dose Group 4; SRD: Dose Group 1; SRD: Dose Group 2; SRD: Dose Group 3
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The main objectives of this trial are to investigate safety, tolerability and pharmacokinetics (PK) of BI 1291583 in healthy male Japanese subjects following oral administration of single rising doses and multiple doses.

ELIGIBILITY:
Inclusion criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests at screening visit
* Japanese ethnicity, according to the following criteria: born in Japan, have lived outside of Japan <10 years, and have parents and grandparents who are Japanese
* Age of 20 to 45 years (inclusive) at screening visit
* BMI of 18.5 to 25.0 kilograms divided by height in meters squared (kg/m2) (inclusive) at screening visit
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation
* Subjects who agree to minimize the risk of making their partner pregnant by fulfilling any of the following criteria starting from the first administration of trial medication until 90 days after last administration of trial medication

  * Use of adequate contraception, any of the following methods plus condom: intrauterine device, combined oral contraceptives that started at least 2 months prior to the first drug administration
  * Vasectomized (vasectomy at least 1 year prior to enrolment)
  * Surgical sterilization (including bilateral tubal occlusion, hysterectomy or bilateral oophorectomy) of the subject's female partner

Exclusion criteria:

* Any finding in the medical examination (including BP, PR, or ECG) deviating from normal and assessed as clinically relevant by the investigator at screening visit
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm) at screening visit
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance at screening visit
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator

  * Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, or hormonal disorders
  * Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
  * Chronic or relevant acute infections including viral hepatitis human immunodeficiency virus (HIV) and/or syphilis
* History of cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days of planned administration of trial medication that might reasonably influence the results of the trial (including drugs that cause QT / QTc interval prolongation [QT: Time between start of the Q-wave and the end of the T-wave in an electrocardiogram, QTc: QT interval corrected for heart rate using the method of Fridericia (QTcF) or Bazett (QTcB)]
* Futher exclusion criteria apply

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-02-04 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
Occurrence of any treatment-emergent adverse event assessed as drug-related by the investigator | up to 65 days

SECONDARY OUTCOMES:
SRD: Area under the concentration-time curve of BI 1291583 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | up to 29 days
  SRD: single-rising dose
SRD: Maximum measured concentration of BI 1291583 in plasma (Cmax) | up to 29 days
  SRD: single-rising dose
MD: After the first dose: Area under the concentration-time curve of BI 1291583 in plasma over a uniform dosing interval τ (AUCτ,1) | up to 24 hours
  MD: multiple doses
MD: After the first dose: Maximum measured concentration of BI 1291583 in plasma (Cmax,1) | up to 24 hours
  MD: multiple doses
MD: After the last dose: Area under the concentration-time curve of BI 1291583 in plasma at steady state over a uniform dosing interval τ (AUCτ,ss) | at day 28
  MD: multiple doses
MD: After the last dose: Maximum measured concentration of BI 1291583 in plasma at steady state (Cmax,ss) | at day 28
  MD: multiple doses

CONTACTS AND LOCATIONS:
Locations (1):
- SOUSEIKAI Sumida Hospital, Tokyo, Sumida-ku, Japan

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com/